CLINICAL TRIAL: NCT03113071
Title: A Phase Ib/II Study of the Safety and Activity of Digoxin With Decitabine in Adult AML and MDS
Brief Title: Safety and Activity of Digoxin With Decitabine in Adult AML and MDS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1061; HM-091 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Decitabine; Digoxin

STUDY DESIGN:
Intervention Model Description: For Group#1 a total of 37 patients with newly diagnosed MDL or MDS will be enrolled, including the eligible patients originally enrolled in the phase Ib portion (safe dose group) of the study, with the goal of determining the clinical activity of our experimental regimen. In the phase II segment, all new patients who are enrolled will initially be randomized in a 1 to 1 fashion to receive decitabine alone or decitabine plus digoxin for one cycle before receiving decitabine plus digoxin for all subsequent cycles for a total of 6 cycles.
  For Group#2 the target will be to enroll a total of 60 patients with relapsed or refractory AML/MDS, including the eligible patients enrolled in the phase Ib group. This group will have randomization and treatments similar to Group#1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Newly diagnosed AML/MDS (Experimental): For Group#1 a total of 37 patients with newly diagnosed MDL or MDS will be enrolled, including the eligible patients originally enrolled in the phase Ib portion (safe dose group) of the study, with the goal of determining the clinical activity of our experimental regimen. In the phase II segment, all new patients who are enrolled will initially be randomized in a 1 to 1 fashion to receive decitabine alone or decitabine plus digoxin for one cycle before receiving decitabine plus digoxin for all subsequent cycles for a total of 6 cycles.
  Interventions: Drug: Decitabine; Drug: Digoxin
- Refractory or relapsed AML/MDS (Experimental): or Group#2 the target will be to enroll a total of 60 patients with relapsed or refractory AML/MDS, including the eligible patients enrolled in the phase Ib group. This group will have randomization and treatments similar to Group#1.
  Interventions: Drug: Decitabine; Drug: Digoxin

INTERVENTIONS:
Drug: Decitabine — Decitabine will be administered in combination with Digoxin
Drug: Digoxin — Decitabine will be administered in combination with Digoxin

SUMMARY:
The primary hypothesis is that digoxin can be safely added to decitabine and will increase the response rates in medically unfit patients with newly diagnosed AML/MDS or those with relapsed/refractory AML/MDS. Furthermore, it is hypothesized that the addition of digoxin to decitabine will result in distinct epigenetic alterations in AML/MDS patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a confirmed diagnosis of one of the following:

   * Newly diagnosed AML (excluding APL)
   * Newly diagnosed intermediate-2 (INT-2) or high-risk MDS
   * Relapsed or Refractory AML, or INT-2 or high-risk MDS
2. For patients with refractory disease they must be at least 4 weeks out from most recent therapeutic intervention.
3. Age > 18 years.
4. ECOG performance status 0 - 2.
5. Patients must have normal organ function as defined below:

   * Total bilirubin within normal institutional limits
   * AST/ALT (SGOT/SGPT) < 2 times institutional normal limits
   * Creatinine within normal institutional limits OR
   * Creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
6. Ability to understand and willingness to sign a written informed consent and HIPAA consent document.
7. Agreement on the part of any male participant to use effective contraception during sexual activity throughout the duration of treatment and for 2 months after discontinuation, for protection against the risk of embryofetal toxicity.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events (less than or equal to Grade 1 toxicity) due to agents administered more than 4 weeks earlier.
2. Patients receiving any other investigational agents.
3. Patients with known brain metastases, active infection, or untreated CNS leukemia.
4. Patients with prior or current history of digoxin exposure.
5. Patients requiring treatment with one or more medications known to interact adversely with digoxin, namely thiazide and/or loop diuretics, quinidine, ritonavir, amiodarone, cyclosporine, itraconazole, propafenone, spironolactone, verapamil.
6. Patients requiring treatment with one or more beta-blockers (metoprolol, atenolol, propranolol) or calcium channel blockers with AV-nodal blocking activity (verapamil, diltiazem).
7. Patient with history of prior exposure to decitabine.
8. Patients eligible for intensive induction chemotherapy and "Medically unfit" based on a TRM score ≥ 13.1*

   * TRM Score= A scoring model which predicts early death following intensive induction chemotherapy in newly diagnosed AML.

     * Model looks at ECOG PS, Age, Platelet Count, Albumin, 2nd AML, WBC, % Peripheral Blasts, Creatinine
     * Score above 13.1 associated with 31%+ chance of death after induction
9. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
10. Known HIV-positive patients on combination anti-retroviral therapy are ineligible because of the potential for pharmacokinetic interactions with digoxin. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
11. Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2019-01-08 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jeans Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Newly Diagnosed AML/MDS | Refractory or Relapsed AML/MDS
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: No patients accrued to Refractory or relapsed AML/MDS arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Newly Diagnosed AML/MDS | Refractory or Relapsed AML/MDS | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Digoxin in Combination With Standard Dose of Decitabine in Patients Newly Diagnosed AML/MDS or Those With Relapsed or Refractory AML/MDS Considered Unfit for Induction Therapy
Description: Maximum tolerated dose of digoxin in combination with standard dose of decitabine will be determined by a standard 3+3 dose de-escalation design
Time Frame: 1-2 months
Population: No patients analyzed because no patients underwent protocol treatment
Arm/Group | Newly Diagnosed AML/MDS | Refractory or Relapsed AML/MDS
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Grade II and IV Toxicities Due to of the Combination Therapy of Decitabine in Combination With Digoxin
Description: The safety of the combination therapy will be determined by the number of grade III or IV non-hematologic toxicities as per NCI CTCAE v4.03 criteria.
Time Frame: 1-3 years
Population: No patients analyzed because no patients underwent protocol treatment
Arm/Group | Newly Diagnosed AML/MDS | Refractory or Relapsed AML/MDS
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Number of MDS Patients With Complete Remission (CR)
Description: Complete response will be assessed by International Working Group (IWG) criteria for MDS
Time Frame: 1-3 years
Population: No patients analyzed because no patients underwent protocol treatment
Arm/Group | Newly Diagnosed AML/MDS | Refractory or Relapsed AML/MDS
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Number of AML Patients With Complete Remission With Incomplete Blood Count Recovery (CRi)
Description: CRi will be assessed by IWG criteria for AML
Time Frame: 1-3 years
Population: No patients analyzed because no patients underwent protocol treatment
Arm/Group | Newly Diagnosed AML/MDS | Refractory or Relapsed AML/MDS
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Description: Adverse event data was not collected because no patients underwent protocol treatment
Arm/Group | Newly Diagnosed AML/MDS | Refractory or Relapsed AML/MDS
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT03113071/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT03113071/ICF_001.pdf